CLINICAL TRIAL: NCT04512651
Title: The Effect of the Thrust Technique of Tibiotarsal Joint on the Symptomatology of Pain at Classical Ballet Dancers
Brief Title: The Thrust Technique of Tibiotarsal Joint on the Symptomatology of Pain at Classical Ballet Dancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do PiauÍ (Other)
Responsible Party: Principal Investigator, Laiana Sepúlveda de Andrade Mesquita, Responsible Researcher, Universidade Estadual do PiauÍ
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2.064.502
Record Dates: First submitted 2020-08-08; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Pain; Osteopathia; Ankle Injuries
Keywords: Osteopathy; Thrust; Classical Ballet; Pain
MeSH Terms: conditions — Pain; Bone Diseases; Ankle Injuries

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial of quantitative character.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): The GI dancers, submitted to tibiotarsal thrust manipulation
  Interventions: Other: Tibiotarsal Thrust Manipulation
- Control Group (CG) (Sham Comparator): For the CG was performed the simulation of the technique, with the participants and the osteopath positioned in the same way as the IG, however there was no reproduction of joint noise.
  Interventions: Other: Simulation Tibiotarsal Thrust Manipulation

INTERVENTIONS:
Other: Tibiotarsal Thrust Manipulation — The dancers were positioned in dorsal decubitus position with the heel outside the stretcher. The osteopath positioned in a lateral feint, inflected knees and forearms in the same plane as the participant's leg. With the internal hand slipped the pinky finger on the medial edge of the foot to the talus neck, the other fingers on the dorsum of the foot and the thumbs controlling the first metatarsus. The position of the talus in relation to the tibia was corrected, initially by placing the foot in eversion and then in dorsal flexion. The osteopath left the body weight behind, causing a traction in the joint. The thrust consisted of a impulse of high speed and low amplitude impulse in a caudal direction, closing the elbows20. The technique was performed until the obtainment (achieved) the joint noise only in the restricted foot, and only one service was performed. After one week, a reassessment of the painful sensation after the dance was performed.
  Arms: Intervention Group (IG)
Other: Simulation Tibiotarsal Thrust Manipulation — Simulation of the technique Tibiotarsal Thrust Manipulation, with the participants and the osteopath positioned in the same way as the IG, however there was no reproduction of joint noise.
  Arms: Control Group (CG)

SUMMARY:
Classical ballet is a type of high performance dance that requires great effort and extreme joint positions by its dancers, not to mention a precise control of the ankle joint when on pointe position. Ballet dancers excessively dorsiflex, and especially plantar flex the ankle, which predisposes anterior displacement of the talus, possibly causing mobility restrictions of the tibiotarsal articulation and making it difficult and painful to move the ankle while dancing. The Thrust technique of tibiotarsal joint is a manipulation that aim to improve mobility and articular function through a high-speed and short-range movement. The purpose of the study is to verify the effect of the Thrust technique of tibiotarsal joint on the pain symptomatology in classical ballet dancers. Ballerinas included in the study presented pain in the ankle when dancing classical ballet, tenderness to palpation in the anterior and posterior tibiotarsal articulation, and dysfunction after compression of the tibiotarsal articulation. The sample consisted of 20 ballerinas, out of which 10 were subjected to manipulation (IG) and 10 formed the control group (CG). Algic symptomatology in classical ballet dance was assessed after some practice with the Visual Analogue Scale (VAS). After that, an algometer was used to quantify the threshold of pain in the anterior and posterior ankle joint that presented restrictions in mobility. The Tug technique was performed in the tibiotarsal articulation in the IG, and in the CG it was simulated. The threshold of pain in the anterior and posterior tibiotalar joint was measured again immediately after the intervention or simulation. The ballerinas were reassessed using algometry and the Visual Analogue Scale (VAS) one week after the manipulation.

DETAILED DESCRIPTION:
This is a randomized clinical trial of quantitative character, realized in a classical ballet school in Teresina, Piauí, Brazil, from June to October 2017. The present research was approved by the Ethics and Research Committee of State University of Piauí. The participants or their guardians signed the Term of Free and Informed Consent in accordance with Resolution 466/12 of the National Health Council (CNS).

The Random randomization in two groups (n=10, each) happens through drawing lots, with the intervention group (GI) submitted to the thrust technique of the tibiotarsal joint for decoaptation of this joint, and the control group (GC), to its simulation.

The instruments used to data collect from the study were: (1) Visual Analog Scale (VAS), a scale that quantifies the intensity of pain through punctuated values, at one extreme of 0, indicating "no pain", to 10, pointing an "maximum pain" 19; (2) Digital algometer (Wagner Instuments®) with a capacity of ten kilograms-force (kgf) and compression deformation of 10 cm, to evaluate the threshold of painful pressure; (3) Questionnaire, developed by the researchers, relating to personal and anthropometric data and related to the ballet practice.

The data collection was carried out in an evaluation room at the ballet school, after the dancers had participated of the classical dance, by a research assistant that was blind to conditions for treatment. The evaluation of the dysfunction in compression of tibiotarsis and the osteopathic manipulation were performed by an experienced osteopath and familiarized with the technique.

To determine the presence of tibiotarsal compression dysfunction in dancers who presented pain during dancing and on palpation at the anterior and posterior tibiotalar joint, the tibiotarsal coaptation and decoaptation test was performed20 (Figure 01): the participants were positioned in dorsal decubitus, already the osteopath, with the internal hand slipped the pinky finger on the medial edge of the foot to the talus neck, the other fingers on the dorsum of the foot and the thumbs on the sole of the foot, the ankle of the dancer was kept in slight inversion and plantar flexion, the therapist flexed his knees, until his forearms stay in the same level as the lower limbs of the participant. Shortly after tractioned and related the joint to perceive if there articulation mobility, or if the joint was fixed.

The VAS was used to weighting (evaluate) the effects on pre and post-test of the osteopathic manipulation, and the algometer checked quantitatively. The points measured by this instrument were the anterior and posterior tibiotalar joint. Before the evaluation, the dancers were submitted to familiarity with the equipment in the triceps surae, in which they were orientated to inform when the pressure would become a painful sensation. In the assessment, the algometer was positioned perpendicularly at the aforementioned points (Figure 01).

The GI dancers, submitted to tibiotarsal thrust manipulation (Figure 02), were positioned in dorsal decubitus position with the heel outside the stretcher. The osteopath positioned in a lateral feint, inflected knees and forearms in the same plane as the participant's leg. With the internal hand slipped the pinky finger on the medial edge of the foot to the talus neck, the other fingers on the dorsum of the foot and the thumbs controlling the first metatarsus. The position of the talus in relation to the tibia was corrected, initially by placing the foot in eversion and then in dorsal flexion. The osteopath left the body weight behind, causing a traction in the joint. The thrust consisted of a impulse of high speed and low amplitude impulse in a caudal direction, closing the elbows20. The technique was performed until the obtainment (achieved) the joint noise only in the restricted foot, and only one service was performed. After one week, a reassessment of the painful sensation after the dance was performed.

For the CG was performed the simulation of the technique, with the participants and the osteopath positioned in the same way as the IG, however there was no reproduction of joint noise.

ELIGIBILITY:
Inclusion Criteria:

Classical ballet dancers with a minimum period of 02 years of practice and who presented pain complaints in the ankle during ballet training, pain at palpation in the anterior and posterior tibiotalar joint of the ankle and dysfunction in compression of the tibiotarsal joint.

Exclusion Criteria:

* Classical ballet dancers with joint hypermobility, painful symptomatology without tibiotarsal compression of the dysfunction and participants who suffered some injury during the survey period.

Ages: 15 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | One week
  A scale that quantifies the intensity of pain through punctuated values, at one extreme of 0, indicating "no pain", to 10, pointing an "maximum pain"

CONTACTS AND LOCATIONS:
Locations (1):
- Laiana Sepúlveda de Andrade Mesquita, Teresina, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No